CLINICAL TRIAL: NCT04174391
Title: Lifestyles for the Prevention of Relapses Among Women with Early Breast Cancer
Brief Title: Lifestyles and Breast Cancer
Acronym: LifeBreast
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Navarra (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Estefania Toledo, Full Professor, University of Navarra
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2019.046
Record Dates: First submitted 2019-11-15; First posted 2019-11-22 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Malignant Tumor of Breast
Keywords: breast cancer prognosis; Mediterranean diet; extra-virgin olive oil; low-fat diet
MeSH Terms: conditions — Breast Neoplasms | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mediterranean diet supplemented with extra-virgin olive oil (Experimental)
  Interventions: Behavioral: Mediterranean diet supplemented with extra-virgin olive oil
- Low-fat diet (Active Comparator)
  Interventions: Behavioral: Low-fat diet

INTERVENTIONS:
Behavioral: Mediterranean diet supplemented with extra-virgin olive oil — Dietary advice on how to follow a Mediterranean diet will be received by the intervention group. The intervention will be delivered mainly by phone (1 call/month), internet and written materials. Also, there will be yearly face-to-face individual interviews and biannual group sessions. A total of 0.5l/week of EVOO for free will be received by participants of this group. In addition, advice on physical activity will be provided.
  Arms: Mediterranean diet supplemented with extra-virgin olive oil
Behavioral: Low-fat diet — Dietary advice on how to follow a low-fat diet will be received by the intervention group. The intervention will be delivered mainly by phone (1 call/month), internet and written materials. Also, there will be yearly face-to-face individual interviews and biannual group sessions. Allotments of commercial foods - equivalent to the extra-virgin olive oil allotment - will be received by participants of this group for free. In addition, advice on physical activity will be provided.
  Arms: Low-fat diet

SUMMARY:
Background: In Spain, 1 out of every 11 women will have a breast cancer before the age of 85 years and breast cancer is the leading cause of potential years of life lost. The randomized intervention in PREDIMED trail, using Mediterranean diet with free provision of extra virgin olive oil (MedDiet+EVOO) dramatically and significantly reduced the occurrence of cases of postmenopausal breast cancer.

Objectives: Assess the efficacy of a nutritional intervention with MedDiet+EVOO for the prevention of relapses among women with early breast cancer.

Methods: Randomized, multicenter trial (LifeBreast) among 766 women diagnosed with early breast cancer. Participants will be randomized in a 1:1 ratio to i) MedDiet+EVOO or ii) low-fat diet. Changes in circulating tumor cells, inflammatory biomarkers, oxidative stress and quality of life will be evaluated. The intervention will be delivered by face-to-face interviews with study dietitian, phone calls, and online tools. Participants in the MedDiet+EVOO group will receive 0.5l/week of EVOO and participants in the low-fat group will receive allotments of different foods, both at no cost. Generalized estimating equations will be used to estimate between-group differences in the following outcomes: circulating tumor cells, inflammatory biomarkers, oxidative stress, and quality of life will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Women with primary pathologically confirmed invasive breast adenocarcinoma in stages I, II or IIIA

Exclusion Criteria:

* breast cancer recurrence
* in situ CDIS or LDIS
* inability or unwillingness to give written informed consent
* difficulty to comply with the intervention
* lack of willpower to change their diet (using the models of Prochaska and DiClemente)
* inability or unwillingness to communicate with study personnel
* medical condition that prevents the intervention (digestive disease with fat intolerance; severe psychiatric, neurological or endocrine disease; or allergy or hypersensitivity to any of the key foods of the intervention (EVOO or nuts) or impossibility to follow a Mediterranean diet and/or EVOO intake
* immunodeficiency or HIV-positive status
* concomitant condition that limits life-expectancy to less than 1 year
* difficulty or impossibility for an adequate follow-up
* institutionalized patients with lack of autonomy
* impossibility for attending group sessions and yearly follow-up visits or for telephone contact
* usual alcohol consumption >80 g/d
* BMI>40
* Patients with acute infection or inflammatory process (e.g. pneumonia) may be included in the study three months after the resolution of the infectious symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 766 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Presence of circulating tumour cells | average follow-up: 1.5 years and then extended to 3.5 years
  Blood samples will be collected at baseline and yearly thereafter. Presence of circulating tumour cells will be determined with immunohistochemical techniques and defined as ≥1 circulating tumour cell in 10 ml of peripheral blood.
Changes in inflammatory markers | average follow-up: 1.5 years and then extended to 3.5 years
  Changes in the inflammatory profile of the participants as plasma cytokines - such as IL-6 -, changes in oxidative stress response with the lipid peroxidation test (LPO test), and changes in DNA damage with electrophoresis single-cell alkaline (comet Assay) in buffy coat will be assessed.

SECONDARY OUTCOMES:
Changes in quality of life | average follow-up: 1.5 years and then extended to 3.5 years
  Changes in quality of life will be assessed with the 36-Item Short Form Survey (SF-36) questionnaire. The questionnaire score ranges from 0-100, with higher score meaning better outcomes.
Changes in quality of life | average follow-up: 1.5 years and then extended to 3.5 years
  Changes in quality of life will be assessed with the the Functional Assessment of Cancer Therapy - Breast (FACT-B) questionnaire. The questionnaire score ranges from 0-148, with higher score meaning better outcomes.
Changes in body mass-index | average follow-up: 1.5 years and then extended to 3.5 years
  Weight and height will be ascertained at baseline and yearly thereafter Weight and height will be directly measured in triplicate by trained study personnel

OTHER OUTCOMES:
Changes in lipid profile | average follow-up: 1.5 years and then extended to 3.5 years
  Blood samples will be collected at baseline and yearly thereafter. Blood samples will be obtained after an overnight fast to determine levels of cholesterol using standard enzymatic methods.
Changes in lipid profile | average follow-up: 1.5 years and then extended to 3.5 years
  Blood samples will be collected at baseline and yearly thereafter. Blood samples will be obtained after an overnight fast to determine levels of triglycerides using standard enzymatic methods.
Changes in blood glucose | average follow-up: 1.5 years and then extended to 3.5 years
  Blood samples will be collected at baseline and yearly thereafter. Blood samples will be obtained after an overnight fast to determine levels of fasting blood glucose using standard enzymatic methods.
Changes in mammographic density | average follow-up: 1.5 years and then extended to 3.5 years
  All available digital mammograms during follow-up of the contralateral non-affected breast of each woman will be collected, they will be read by an experienced radiologist in a blind way (without knowing the allocation group) using the DM-Scan program.
HOMA-IR and HOMA-beta | average follow-up: 3.5 years
  HOMA-IR and HOMA-beta will be calculated based on serum glucose and insulin concentrations. They will be measured by standard laboratory methods.

CONTACTS AND LOCATIONS:
Overall Officials: Estefania A Toledo, MD, MPH, PhD, Principal Investigator — University of Navarra (IdiSNA); Trinidad Dierssen-Sotos, MD, PhD, Principal Investigator — University of Cantabria; Jose J Jimenez-Moleon, MD, PhD, Principal Investigator — Instituto de Investigación Biosanitaria de Granada (ibs.Granada); Marina Pollan, Md, PhD, Principal Investigator — Instituto de Salud Carlos III
Locations (4):
- Spain (4):
  - University of Cantabria, Santander, Cantabria
  - Instituto de Investigación Biosanitaria de Granada ibs.GRANADA, Granada, Granada
  - University of Jaen, Jaén, Jaen
  - University of Navarra-Instituto de Investigación Sanitaria de Navarra, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: Undecided